CLINICAL TRIAL: NCT03033082
Title: Evaluation of Marital and Sexual Satisfaction of Wives to Erectile Dysfunction Males Using Intra Corporeal Injection (Ici). In Correlation to Personality Profile
Brief Title: Evaluation of Marital and Sexual Satisfaction of Wives to Erectile Dysfunction Males
Status: Completed | Type: Observational
Sponsor: Adam International Hospital (Other)
Responsible Party: Principal Investigator, Ahmad Raef Sadek, Prinicipal Investigator Ahmad Raef, Adam International Hospital
Other Study IDs: 2014
Record Dates: First submitted 2017-01-22; First posted 2017-01-26 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Erectile dysfunction patients: Questionnaire sheets.
  Interventions: Other: Questionnaire sheets
- Normal males: Questionnaire sheets.
  Interventions: Other: Questionnaire sheets

INTERVENTIONS:
Other: Questionnaire sheets — A- Marital satisfaction Index (MSI). Interview (Modified Arabic translation)
  B- Sexual Satisfaction Scale:(SSS). The Arabic version of the sexual satisfaction scale was used.
  C- International Index of Erectile Function Questionnaire (IIEF-5): For male subjects.
  D- The Eysenck Personality Questionnaire (EPQ):
  The Arabic version of the EPQ was used.

SUMMARY:
Erectile Dysfunction (ED), previously known as sexual impotence, is defined as the persistent inability to obtain and/or maintain a penile erection that is hard enough for satisfactory sexual intercourse. The number of reported patients with ED is increasing and it is becoming a real medical problem.

DETAILED DESCRIPTION:
Marital satisfaction is a global evaluation of the state of one's marriage or current long-term romantic relationship. This global evaluation can be a reflection of a how happy people are in their marriage in general or a composite of satisfaction with several specific facets of the marital relationship. Sexual health can be described as enjoying and fulfilling sexual desires without harming, physical or psychological, oneself or others. Sexual functioning is an important part of a patient's health and well-being. Patients often seek for treatment late due to embarrassment and commonly with an alternative problem. Sexual and erectile functions are considered important components of men's overall health. The psychosocial impact of ED can lead to depression, loss of self-esteem, and relationship and marital difficulties. Personality is defined as the "distinctive and characteristic patterns of thought, emotion and behavior that define an individual's personal style and influence his or her interaction with the environment".

ELIGIBILITY:
Inclusion Criteria:

* Married couples

Exclusion Criteria:

* Unmarried couples.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Males complaining of erectile dysfunction.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2014-06-01 (Actual); Study Completion 2014-06-30 (Actual)

PRIMARY OUTCOMES:
Marital and sexual satisfaction. | Six months.
  Questionnaire sheets.

IPD SHARING:
Plan to Share IPD: Yes
Contact the authors